CLINICAL TRIAL: NCT07366645
Title: Clinical Efficacy and Cost-Effectiveness of Silver Diamine Fluoride and Silver Fluoride to Arrest Incipient Carious Lesions in Permanent Molar Teeth With or Without Application of LED Light: A Randomized Clinical Trial
Brief Title: Clinical and Cost-Effectiveness of Silver Diamine Fluoride and Silver Fluoride, With or Without Application of LED, in Arresting Incipient Permament Molar Caries
Acronym: SDF and AgF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Amr Khodair, Lecturer Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3344515
Record Dates: First submitted 2025-12-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Incipient Caries
MeSH Terms: interventions — silver fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Pits and fissures receive International Silver Diamine Fluoride for caries arrest (Active Comparator): Remineralization and prevention of incipient pits and fissure caries of permanent molars by International Silver Diamine Fluoride application for 60 seconds
  Interventions: Other: International Sliver Diamine Fluoride
- Pits and fissures receive Local brand Egyptian Sliver Diamine Fluoride for caries arrest (Experimental): Remineralization and prevention of incipient pits and fissure caries of permanent molars by local brand Egyptian Silver Diamine Fluoride application for 60 seconds
  Interventions: Other: Local brand Egyptian Silver Diamine Fluoride
- Pits and fissures receive Sliver Fluoride for caries arrest (Experimental): Remineralization and prevention of incipient pits and fissure caries of permanent molars by Silver Fluoride application for 60 seconds
  Interventions: Other: Silver Fluoride
- Pits and fissures receive International Silver Diamine Fluoride with LED for caries arrest (Experimental): Remineralization and prevention of incipient pits and fissure caries of permanent molars by Silver Diamine Fluoride application for 10 seconds, followed by the application LED light for 20 seconds
  Interventions: Other: International Sliver Diamine Fluoride with LED light
- Pits and fissures receive local brand Egyptian Silver Diamine Fluoride with LED for caries arrest (Experimental): Remineralization and prevention of incipient pits and fissure caries of permanent molars by local brand Egyptian Silver Diamine Fluoride application for 10 seconds, followed by LED light for 20 seconds
  Interventions: Other: Local brand Egyptian Silver Diamine Fluoride with LED light
- Pits and fissures receive Sliver Fluoride with LED for caries arrest (Experimental): Remineralization and prevention of incipient pits and fissure caries of permanent molars by Silver Fluoride application for 10 seconds, followed by application of LED light for 20 seconds
  Interventions: Other: Silver Fluoride with LED light

INTERVENTIONS:
Other: International Sliver Diamine Fluoride — It is the gold standard; it is an international brand, it is ammonia-based, and it is a remineralizing agent with an application time of 60 seconds.
  Arms: Pits and fissures receive International Silver Diamine Fluoride for caries arrest
Other: Local brand Egyptian Silver Diamine Fluoride — It is a new Egyptian brand of SDF; it is ammonia-based, and it is a remineralizing agent with an application time of 60 seconds.
  Arms: Pits and fissures receive Local brand Egyptian Sliver Diamine Fluoride for caries arrest
Other: Silver Fluoride — It is a water-based remineralizing agent with an application time of 60 seconds.
  Arms: Pits and fissures receive Sliver Fluoride for caries arrest
Other: International Sliver Diamine Fluoride with LED light — It is an international brand, it is ammonia-based, and it is a remineralizing agent with an application time of 10 seconds, followed by LED light application for 20 seconds.
  Arms: Pits and fissures receive International Silver Diamine Fluoride with LED for caries arrest
Other: Local brand Egyptian Silver Diamine Fluoride with LED light — It is a new Egyptian brand of SDF; it is ammonia-based, and it is a remineralizing agent with an application time of 10 seconds, followed by LED application for 20 seconds.
  Arms: Pits and fissures receive local brand Egyptian Silver Diamine Fluoride with LED for caries arrest
Other: Silver Fluoride with LED light — It is a water-based remineralizing agent with an application time of 10 seconds, followed by LED light application for 20 seconds.
  Arms: Pits and fissures receive Sliver Fluoride with LED for caries arrest

SUMMARY:
The study aims to compare the effect of international brand ammonia based 38% SDF, water based silver fluoride solution (AgF), an aqueous silver fluoride solution, and local brand ammonia based SDF with and without LED light application on caries arrest of initial enamel pits and fissure caries for permanent teeth of young adults

ELIGIBILITY:
Inclusion Criteria:

* high caries risk dental students
* Males or females
* Medically free
* Not taking medication
* At least had one active carious tooth
* Posterior permanent teeth
* ICDAS 2

Exclusion Criteria:

* non-Egyptian students
* Lack of compliance
* Allergic reaction to the materials used
* Pregnancy
* Dental students cannot give consent
* Teeth that will be extracted for orthodontic reasons
* Dental fluorosis
* Hypo calcified teeth
* Systemic diseases affecting teeth, such as amelogenesis imperfecta
* Severe periodontal affection

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 366 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Caries arrest | After 3, 6, and 12 months.
  Lesion activity will be assessed by caries status (active/inactive) using visual and tactile inspection for surface discontinuities and texture. The participants will be examined under unit light using a 0.5 mm ball-ended (CPI) probe and a dental mirror. The teeth will be cleaned and dried by a water-air spray syringe before the examination.